CLINICAL TRIAL: NCT06728943
Title: Efficacy of Intra-Ureteric Aminophylline Installation After Failed Stone Accessibility by Semi-rigid Ureteroscopy. Prospective Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Fawzy Abd Elfattah Salman, lecturer of urology, Al-Azhar University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Intra-Ureteric Aminophylline
Record Dates: First submitted 2024-12-08; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Ureterocopic Lithotripsy; Stone Ureter; Ureteric Stone
Keywords: ureteroscopy; stone ureter; ureteral dilatation; failed ureteroscopy
MeSH Terms: conditions — Ureterolithiasis

STUDY DESIGN:
Intervention Model Description: Direct semi-rigid ureteroscopy will initially be attempted without endodilatation (KARL STORZ, 43 cm, 6°, 7 Fr.). On failure to advance the semi-rigid ureteroscope through the ureter, intra-ureteric instillation of 20 ml of aminophylline (250 mg/10 mL) through ureteric stent and another trial to pass the same scope will be done after 10 minutes of intra-ureteral aminophylline instillation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The group of patients with failed stone accessibility by semi-rigid ureteroscopy (Experimental): Direct semi-rigid ureteroscopy will initially be attempted without endodilatation (KARL STORZ, 43 cm, 6°, 7 Fr.). On failure to advance the semi-rigid ureteroscope through the ureter, intra-ureteric instillation of 20 ml of aminophylline (250 mg/10 mL) through ureteric stent and another trial to pass the same scope will be done after 10 minutes of intra-ureteral aminophylline instillation.
  Interventions: Procedure: ureteral dilatation

INTERVENTIONS:
Procedure: ureteral dilatation — Direct semi-rigid ureteroscopy will initially be attempted without endodilatation (KARL STORZ, 43 cm, 6°, 7 Fr.). On failure to advance the semi-rigid ureteroscope through the ureter, intra-ureteric instillation of 20 ml of aminophylline (250 mg/10 mL) through ureteric stent and another trial to pass the same scope will be done after 10 minutes of intra-ureteral aminophylline instillation.

SUMMARY:
In this study we will test the effect of local intraureteric aminophylline instillation through Ureteric stent and Reaching stone without the need of ballon dilataion

DETAILED DESCRIPTION:
Urolithiasis is a significantly common disease globally, despite the notable difference in the rate of occurrence based on various factors like gender, climate, diet, and other risk factors. There has been a yearly increase in the prevalence of stone occurrence in people above the age of 30 for all genders. (1).

The EAU recommends URS as the first-line treatment for stones either in the proximal or distal ureter measuring >10 mm; for <10 mm, either URS or SWL can be selected for first-line management. URS is associated with a higher SFR and a better clinical outcome when compared to SWL (1,6.7.8) .

During ureteroscopy, the use of guide wire and ureteroscope itself in the procedures can lead to complications like ureteral spasm. Agents like lidocaine gel, intravenous buscopan and aminophylline can be used to relieve spasm and increase the success of treatment. Aminophylline is used for the treatment of acute phase of renal colic. (2) .

Aminophylline, a methyl xanthine and theophylline derivative, relaxes smooth muscle by increasing the concentration of intracellular 3",5"-cyclic adenosine monophosphate (cAMP), and cyclic guanosine mono- phosphate (cGMP) and activating protein kinase A. In addition, aminophylline alleviates inflammation by decreasing the production of leukotrienes and TNFα. (3) .

Aminophylline is a drug having combination of theophylline and ethylenediamine in a ratio of 2:1. Theophylline helps in peristalsis of ureter and verapamil causes an acute dilation of proximal ureter. The capability to alter the diameter of ureter and the peristaltic activity helps in ureteroscopy. Aminophylline is a cheap, safe, with minimum side effects. (3) .

In a randomized controlled trial, performed by (Shabayek et al., 2022) on the effect of intravesical aminophylline instillation after failure of advancing semi-rigid ureteroscope through the ureteric orifice without endodilatation. Intravesical aminophylline instillation was effective in reducing intraureteral pressure at the lower ureter and can be used as an alternative to balloon dilatation prior to ureteroscopic management of distal ureteric stones.

In a study performed by (Lubana et al., 2024), The use of local aminophylline during ureteroscopic stone treatment has been found to be highly useful and effective in reducing the need of stents and secondary surgery, decreased pain, and increased success rate.

In this study we will test the effect of local intraureteric aminophylline instillation through Ureteric stent and Reaching stone without the need of ballon dilataion

ELIGIBILITY:
Inclusion Criteria:

* The study will include patients with failed stone accessibility by semi-rigid ureteroscopy.

Exclusion Criteria:

* Child age group
* Pre stented patients
* Contraindications to aminophylline (hypersensitivity to drug components, pregnancy or lactation ,…)
* Contraindications to ureteroscopy (active urinary tract infection - Contraindications to general or spinal anesthesia - Uncorrected bleeding disorders)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Success rate of Ureteral access and Scoping of the stones after Intra-ureteral instillation of Aminophylline without Ballon Dilatation | from the start of ureteroscopy entrance to the end of the procedure
  Success rate of Ureteral access and Scoping of the stones after Intra-ureteral instillation of Aminophylline without Ballon Dilatation

SECONDARY OUTCOMES:
Success of complete extraction of stones | from the start of ureteroscopic entrance to the end of the procedure
  Success of complete extraction of stones after intraureteric injection of aminophylline

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar university, faculty of medicine, the urology department, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided